CLINICAL TRIAL: NCT04316741
Title: Harnessing Social Media to Reduce Cannabis Use Among Adolescents and Emerging Adults in an Urban Emergency Department
Brief Title: Brief Intervention Combined With Health Coaching Via Social Media for Cannabis Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00139068; R34DA045712 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Cannabis Use

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention+Health Coaching (Experimental): Brief intervention with social-media delivered health coaching
  Interventions: Behavioral: Snapcoach
- Control (No Intervention): Enhanced usual care brochure plus attention control with social media messaging

INTERVENTIONS:
Behavioral: Snapcoach — A brief motivational interviewing-based intervention combined with health coaching via social media for 4 weeks
  Arms: Brief Intervention+Health Coaching

SUMMARY:
The purpose of the study is to develop and test social media interventions to help young people increase well-being and reduce risky behaviors. The study will help researchers learn about ways to deliver wellness information in a way that is appealing and helpful to young people who use Snapchat.

ELIGIBILITY:
Inclusion Criteria:

Individuals seen in the Emergency Department at Hurley Medical Center who meet these criteria

* self-report of weekly or more frequent cannabis use for past 3 months
* past month Snapchat use
* ability to consent
* English-speaking
* between ages 18-25
* smart phone ownership

Exclusion Criteria:

* Emergency Department presentation for suicidality and/or acute psychosis, being in police custody, or present with psychological distress requiring intensive social work (e.g. sexual assault)
* having a medical cannabis card

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bonar, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred October 2020 through November 2021 with patients who were attending the Emergency Department or had a recent Emergency Department visit.
Pre-assignment Details: N = 63 consented at baseline for the RCT, but 5 were lost to follow-up prior to randomization.
Period: Baseline Enrollment
Arm/Group | Brief Intervention+Health Coaching | Control
Started | 30 | 28
Completed | 29 (29 participants completed some part of the intervention/health coaching) | 27
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Immediate Post-Test
Arm/Group | Brief Intervention+Health Coaching | Control
Started | 29 | 27
Completed | 24 | 26
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1
Period: 1-month Post-test
Arm/Group | Brief Intervention+Health Coaching | Control
Started | 29 | 27
Completed | 22 | 25
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 2
Period: 3-month Follow-up
Arm/Group | Brief Intervention+Health Coaching | Control
Started | 29 | 27
Completed | 19 | 25
Not Completed | 10 | 2
Not completed — Lost to Follow-up | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Intervention+Health Coaching | Control | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (2.4) | 21.8 (2.5) | 21.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 11 | 28
  White | 8 | 10 | 18
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brief Intervention Acceptability
Description: Acceptability rating completed by participants for the brief intervention session
Time Frame: Immediate post-test administered after the session
Population: These data were not collected from the participants in the "Control" Arm/Group. These data refer to the intervention only.
  24 participants who completed ratings of the intervention session immediately post-intervention.
  Acceptability measured by the following item: How much did you enjoy talking to your health coach today?
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention+Health Coaching
Number analyzed (Participants) | 24
Participants
  Liked it/Liked it a lot | 23
  Neutral | 1
  Disliked it/disliked it a lot | 0

2. Primary Outcome: Snapchat Acceptability Rating
Description: Acceptability rating completed by participants for the Snapchat-delivered health coaching.
  Item: In general, I enjoyed the Snapchat messages from the SnapCoach team. (Not at all, A little, Somewhat, Very, Extremely)
Time Frame: 1 month
Population: These data were not collected from the participants in the "Control" Arm/Group. These data refer to the intervention only.
  22 participants in intervention condition who completed a post-test at 1-month after enrollment (i.e., conclusion of intervention period)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention+Health Coaching
Number analyzed (Participants) | 22
Participants
  Not at all | 0
  A little/somewhat | 4
  Very much/extremely | 18

3. Primary Outcome: Brief Intervention Feasibility
Description: % of participants assigned to condition who complete the brief intervention
Time Frame: Immediate
Population: Individuals randomized to intervention condition These data were not collected from the participants in the "Control" Arm/Group. These data refer to the intervention only.
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention+Health Coaching
Number analyzed (Participants) | 30
Participants
  completed brief intervention session | 26
  did not complete brief intervention session | 4

4. Primary Outcome: Snapchat Health Coaching Feasibility
Description: % of participants who complete key activities (e.g., % who add health coach on Snapchat)
Time Frame: Up to 1 month
Population: 30 individuals randomized to the intervention group These data were not collected from the participants in the "Control" Arm/Group. These data refer to the intervention only.
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention+Health Coaching
Number analyzed (Participants) | 30
Participants
  % who added coaches on Snapchat | 29
  % who did not add coaches on Snapchat | 1

5. Primary Outcome: Snapchat Health Coaching Feasibility
Description: % of participants who complete key activities (e.g., % who reply to at least 1 Snapchat message)
Time Frame: Up to 1 month
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention+Health Coaching
Number analyzed (Participants) | 30
Participants
  % who replied to at least 1 Snapchat message | 26
  % who did not reply to at least 1 Snapchat message | 4

ADVERSE EVENTS:
Time Frame: From baseline enrollment to 3-month follow-up.
Description: Adverse events were standard as for behavioral studies and could include deaths, hospitalizations, etc.
Arm/Group | Brief Intervention+Health Coaching | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

LIMITATIONS AND CAVEATS:
This work occurred in the COVID-19 pandemic ina front-line clinical setting (Emergency Department in an socio-economically under-resourced community). COVID-related shutdowns of in-person research, COVID protocols (e.g., inability to approach participants in droplet precautions), and staffing retention (e.g., abiltiy to employ individuals who would work in a COVID frontline setting) impeded recruitment of the originally planned sample size, with impacts also on retention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04316741/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT04316741/ICF_002.pdf